CLINICAL TRIAL: NCT06776783
Title: A Randomized, Controlled, Blinded, Parallel Group Study of the Safety and Efficacy of APC-0101 (SF-RI 1 Surfactant for Inhalation Combined With a Dedicated Delivery System) in Preterm Infants With Respiratory Distress Syndrome
Brief Title: Safety and Efficacy of APC-0101 in Preterm Infants With Respiratory Distress Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aerogen Pharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APC-AF-CLN-003
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Distress Syndrome; Pre-term Infants
Keywords: respiratory distress syndrome; surfactant; pre-term infant
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding/masking will be accomplished by a two-level redundant process. First, a screen (or private room) will be placed around the subject's bedside area and the APC-0101 Controller during APC-0101 or Sham treatment. This will ensure that no members of the clinical team, other than the blinded bedside nurse, will see the subject or the Controller throughout treatment. Second, the Controller and subject's face will be shielded so the blinded bedside nurse cannot determine whether the subject is receiving APC-0101 or Sham treatment.
  A trained, unblinded, staff member (e.g., a respiratory therapist) will set up the Controller, but will not be involved with making decisions about the respiratory support of the subject.
  Parents and all members of the clinical team who will make decisions about respiratory support, including FiO2, assessment of Failure Criteria, or assessment of AEs, will remain blinded throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control Group (Sham Comparator)
  Interventions: Other: Control
- APC-0101 Group (Experimental)
  Interventions: Combination Product: APC-0101 (SF-RI 1 surfactant for inhalation combined with a dedicated delivery system)

INTERVENTIONS:
Combination Product: APC-0101 (SF-RI 1 surfactant for inhalation combined with a dedicated delivery system) — Subjects in the APC-0101 group will be changed from their current nCPAP/NIV interface to the APC-0101 nCPAP/NIV interface and APC-0101 treatment will be started.
  Arms: APC-0101 Group
Other: Control — Subjects in the Control group will be changed from their current nCPAP/NIV interface to the APC-0101 nCPAP/NIV interface but an empty vial will be used instead of APC-0101.
  Arms: Control Group

SUMMARY:
This is a 2-part, prospective, randomized, blinded, sham-controlled, multi-center study comparing preterm subjects with RDS who are treated with APC-0101 and nCPAP/NIV to subjects treated with nCPAP/NIV alone (Sham). In Part 1, subjects will be followed until they reach 40 weeks post-menstrual age (PMA) or are discharged from the NICU, whichever comes first. In Part 2, subjects will undergo post-term follow-up through 24 months corrected age.

ELIGIBILITY:
Inclusion Criteria:

1. Inborn at the study site's hospital (i.e., not transferred from another hospital following delivery)
2. Gestational age at birth of 26 through 33 weeks PMA
3. Birth weight appropriate for gestational age (AGA, weight 3rd to 97th percentile on Fenton Growth Curve)
4. Birth weight ≤ 2000 grams
5. Post-natal age 1 to 24 hours at randomization
6. On nCPAP or NIV for at least 30 minutes with RSS = 1.4 - 2.0 to maintain SpO2 90-95% at randomization. RSS is calculated as (nCPAP cm H2O) × (FiO2) or as (NIV mean airway pressure cm H2O) × (FiO2).
7. FiO2 ≥ 0.24 at randomization
8. nCPAP or mPaw ≥ 6 cm H2O at randomization
9. Chest radiograph (CXR) or lung ultrasound compatible with RDS prior to randomization

Exclusion Criteria:

1. On SiPAP®, RAM® cannula, or high flow nasal cannula (HFNC) (> 2 liters per minute [LPM]) at the time of randomization
2. Prior instillation of surfactant
3. Premature rupture of membranes (PROM) occurring > 14 days before birth
4. Significant congenital/chromosomal anomaly (e.g., Pierre Robin syndrome, clinically significant congenital heart disease, or trisomy)
5. Pneumothorax
6. Other etiologies of respiratory distress
7. Enrollment in another interventional study with similar efficacy endpoints
8. Apgar score at 5 min of 0-3
9. Prior cardiopulmonary resuscitation (CPR) or epinephrine
10. Base Deficit > 15 mEq/L on most recent arterial blood gas (not capillary blood gas, venous blood gas, or cord gas) prior to randomization. Note that arterial blood gas is not required prior to randomization.
11. Partial pressure of carbon dioxide (PaCO2) > 65 mmHg on most recent arterial blood gas (not capillary blood gas, venous blood gas, or cord gas) prior to randomization.
12. Triplet or higher order multiple birth

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 520 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Failure Criteria | First 7 days of life
  Number (%) of subjects who meet the predetermined criteria for failure of nCPAP/NIV

SECONDARY OUTCOMES:
Instilled Bolus Surfactant | First 72 hours of life
  The number (%) of subjects in each group who receive instilled bolus surfactant.
Multiple Bolus Surfactant Doses | First 72 hours of life
  The number (%) of subjects in each group who receive multiple doses of bolus surfactant.
Total Number of Bolus Surfactant Doses | First 72 hours of life
  The total number of bolus doses of surfactant received per subject in each group.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UF Health Jacksonville, Jacksonville, Florida
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Goryeb Children's Hospital, Morristown, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Christus Children's Hospital, San Antonio, Texas
  - University of Virginia School of Medicine, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No